CLINICAL TRIAL: NCT00286845
Title: Use of the MiCK Assay for Apoptosis to Predict Complete Remission in Acute Myeloid Leukemia
Brief Title: Use of the MiCK Assay for Apoptosis in AML
Status: Completed | Type: Observational
Sponsor: Pierian Biosciences (Industry)
Collaborators: DiaTech Oncology and Vanderbilt University (Other)
Responsible Party: Cary Presant, MD, DiaTech Oncology
Other Study IDs: Diatech Leuk II Vand
Record Dates: First submitted 2006-01-16; First posted 2006-02-06 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: Chemosensitivity; Acute Myeloid Leukemia; Apoptosis; MiCK Assay
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- II
  Interventions: Drug: Standard Chemotherapy
- 1

INTERVENTIONS:
Drug: Standard Chemotherapy — physician determined
  Groups: II

SUMMARY:
A previous preliminary study performed at Vanderbilt University with funding from the Leukemia Society of America demonstrated that the response of leukemia cells in vitro to the chemotherapeutic agent idarubicin in the microculture kinetic assay for apoptosis (MiCK assay) predicted survival in patients with newly diagnosed acute myeloid leukemia (AML). In this previous study, achievement of complete response (CR) to induction therapy with idarubicin and cytarabine was used as the clinical indicator for determining whether leukemia specimens taken prior to treatment were sensitive or not sensitive in the MiCK assay. This group of patients has been followed for 7 years and their long term survival rates show that their responses in the MiCK assay to idarubicin but not cytarabine predict survival. In the present proposal a separate group of patients with newly diagnosed AML will be recruited to provide leukemia cell samples that will be used to establish criteria for sensitivity and non-sensitivity to idarubicin and cytarabine in the MiCK assay. The achievement of CR will be used to determine in vitro sensitivity as it was done in the previous study. With the in vitro sensitivities as determined in this proposed study, the long term survivals of patients in the previous study will be analyzed prospectively.

The proposed study is expected to have an approximate duration of one year. Patient population will include newly diagnosed AML patients with both de novo AML and AML arising from a previously diagnosed myelodysplastic syndrome. The study will not include patients with previously treated leukemia that has relapsed

DETAILED DESCRIPTION:
A previous preliminary study performed at Vanderbilt University with funding from the Leukemia Society of America demonstrated that the response of leukemia cells in vitro to the chemotherapeutic agent idarubicin in the microculture kinetic assay for apoptosis (MiCK assay) predicted survival in patients with newly diagnosed acute myeloid leukemia (AML). In this previous study, achievement of complete response (CR) to induction therapy with idarubicin and cytarabine was used as the clinical indicator for determining whether leukemia specimens taken prior to treatment were sensitive or not sensitive in the MiCK assay. This group of patients has been followed for 7 years and their long term survival rates show that their responses in the MiCK assay to idarubicin but not cytarabine predict survival. In the present proposal a separate group of patients with newly diagnosed AML will be recruited to provide leukemia cell samples that will be used to establish criteria for sensitivity and non-sensitivity to idarubicin and cytarabine in the MiCK assay. The achievement of CR will be used to determine in vitro sensitivity as it was done in the previous study. With the in vitro sensitivities as determined in this proposed study, the long term survivals of patients in the previous study will be analyzed prospectively.

STUDY DESIGN

1. Recruit patients and assign them unique number at the time of sample collection. All samples and data will be recorded by unique number. The key to the unique numbers assigned to each patient will be kept by the principal investigators at Vanderbilt.
2. After obtaining informed consent, collect specimens from patients whose induction therapy will include cytarabine and idarubicin. Collect and ship to DiaTech by overnight courier fifty (50) bone marrow or peripheral blood [if available, both bone marrow and peripheral blood] specimens from newly diagnosed patients with AML. Newly diagnosed AML patients include those diagnosed de novo or arising from a previously diagnosed myelodysplastic syndrome, but do not include patients with previously treated leukemia that has relapsed. An adequate specimen for analysis will contain sufficient numbers of viable leukemia cells to perform the MiCK assay with 7 doses of cytarabine and 7 doses of idarubicin..
3. Each patient's clinically recognized predictors of leukemia treatment outcome will be recorded. These predictors include age, sex, presence or absence of preceding myelodysplastic syndrome, blood leukocyte count at diagnosis, percentage of leukemic cells in the blood, and leukemic cell karyotype.

ELIGIBILITY:
Inclusion Criteria:

patients with newly diagnosed acute myeloid leukemia (AML

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population will include newly diagnosed AML patients with both de novo AML and AML arising from a previously diagnosed myelodysplastic syndrome. The study will not include patients with previously treated leukemia that has relapsed
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-01; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cary Presant, MD, Principal Investigator — Pierian Biosciences
Locations (1):
- Vanderbilt University Medical Center and DiaTech Oncology, Nashville, Tennessee, United States

REFERENCES:
- [Background] Kravtsov VD. A novel microculture kinetic assay (MiCK assay) for malignant cell growth and chemosensitivity. Eur J Cancer. 1994;30A(10):1564-70. doi: 10.1016/0959-8049(94)00291-c. PMID 7833120
- [Background] Kravtsov VD, Fabian I. Automated monitoring of apoptosis in suspension cell cultures. Lab Invest. 1996 Feb;74(2):557-70. PMID 8780173
- [Background] Kravtsov VD, Greer JP, Whitlock JA, Koury MJ. Use of the microculture kinetic assay of apoptosis to determine chemosensitivities of leukemias. Blood. 1998 Aug 1;92(3):968-80. PMID 9680366
- [Background] Kravtsov VD, Daniel TO, Koury MJ. Comparative analysis of different methodological approaches to the in vitro study of drug-induced apoptosis. Am J Pathol. 1999 Oct;155(4):1327-39. doi: 10.1016/S0002-9440(10)65235-2. PMID 10514415
- [Derived] Strickland SA, Raptis A, Hallquist A, Rutledge J, Chernick M, Perree M, Talbott MS, Presant CA. Correlation of the microculture-kinetic drug-induced apoptosis assay with patient outcomes in initial treatment of adult acute myelocytic leukemia. Leuk Lymphoma. 2013 Mar;54(3):528-34. doi: 10.3109/10428194.2012.722217. Epub 2012 Sep 17. PMID 22924433